CLINICAL TRIAL: NCT05307198
Title: Rectal Artery Infusion Chemotherapy of Oxaliplatin Plus Capecitabine Combined With Anti-PD1 Antibody After Induction Chemotherapy for Microsatellite Stable Locally Advanced Rectal Cancer：a Prospective Single-arm Phase II Study
Brief Title: Rectal Artery Infusion Chemotherapy Combined With Anti-PD1 Antibody for MSS LARC
Acronym: RAIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Jun Li
Record Dates: First submitted 2022-01-10; First posted 2022-04-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-02

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; spartalizumab; sintilimab

STUDY DESIGN:
Intervention Model Description: The pCR rate of neoadjuvant chemoradiotherapy is about 20% (null hypothesis). Assuming that the pCR of the RAIC scheme in this study would be in the range of 15%-35%. Using Simon's two-stage design, a total of 37 patients would provide 80% power at a one sided 5% alpha level. Considering the drop rate of 10%, 38 patients would be included (64 cases to be screened) in this study. 10 cases (17 cases were screened) and 28 cases (47 cases were screened) would be included in the first and second stages, respectively. If the number of patients with pCR in the first stage is less than 2, the study will be terminated. If the number of patients with pCR in the first stage is more than 2, a second-stage trial will be performed. If the total number of patients with pCR is more than 9, the effective remission rate of the RAIC regimen is considered to be acceptable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rectal Artery Infusion Chemotherapy (Experimental): Patients receive 2 cycles of Capecitabine and Oxaliplatin (CapeOx) chemotherapy and evaluated with rectum Magnetic Resonance Imaging (MRI). Patients with more than 20% regression of maximum diameter of rectal tumor in MRI image will entry into next step of rectal artery infusion of Oxaliplatin and oral Capecitabine（1000mg/㎡）with anti-PD1 antibody（200mg）every 3 weeks for 2 cycles.Then those patients will receive rectectomy including anterior resection or abdominoperineal resection by open or laparoscopy with TME.
  Interventions: Drug: Oxaliplatin; Procedure: Rectectomy; Drug: Capecitabine; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Oxaliplatin — Drug: Oxaliplatin Oxaliplatin 130mg/m2 for inducing chemotherapy in Day 1 every 3 weeks and repeat for two cycles.
  The dose of oxaliplatin used for rectal artery infusion was uncertain because there were no previous study. We design this study with Oxaliplatin 85mg/㎡for rectal artery infusion chemotherapy in Day 1 every 3 weeks and repeat for 2 cycles, based on intravenous chemotherapy regimens recommended by NCCN（mFolfox6）.If there were severe side effects caused by oxaliplatin observed within first 5 patients, we would decreasing the dose of oxaliplatin depending on the multidisciplinary discussion of researchers.
  We acknowledged that our study did not determine the most appropriate dosage of oxaliplatin used for artery infusion, but rather performed a novel therapeutic method for microsatellite stable locally advanced rectal cancer.
Procedure: Rectectomy — Include anterior resection or abdominoperineal resection by open or laparoscopy with Total Mesorectal Excision (TME).
Drug: Capecitabine — Oral Capecitabine 1000 mg/m2 twice daily combined with oxaliplatin chemotherapy in Day 1 to Day 14 every 3 weeks and repeat for 4 cycles.
Drug: Anti-PD-1 monoclonal antibody — Anti-PD1 antibody 200mg/m2 in Day 2 after Rectal Artery Infusion Chemotherapy. Repeat every 3 weeks for 2 cycles.
  Other Names: Sintilimab

SUMMARY:
The purpose of this study is to explore whether rectal artery infusion chemotherapy combined with anti-PD1 antibody is an effective neoadjuvant therapy for the microsatellite stable locally advanced rectal cancer.

DETAILED DESCRIPTION:
Neoadjuvant chemoradiation is the standard treatment for locally advanced rectal cancer. Neoadjuvant chemoradiotherapy can achieve a pathological complete response rate (pCR) of about 20%. However, radiotherapy can cause tissue edema and fibrosis, increasing the risk of anastomotic leakage, resulting in rectal, urinary, and sexual dysfunction. Neoadjuvant chemotherapy or immunotherapy can avoid these adverse reactions, but the pCR rate of chemotherapy is significantly lower than that of neoadjuvant radiotherapy, and immunotherapy is less effective for MSS patients with weak immunogenicity. This study is a prospective, single-arm, single-center trial. The study will enhance the local killing effect of oxaliplatin through rectal artery infusion and induce immunogenic cell death (ICD) to enhance tumor antigen presentation, and then combine anti-PD1 antibody for neoadjuvant therapy. The study will address whether this treatment combination achieves pCR rates that are non-inferior to neoadjuvant RT for MSS-type locally advanced rectal cancer. It is known that the effective rate of oxaliplatin-containing intravenous chemotherapy for colorectal cancer is about 60%. In this study, 2 cycles of XELOX induction chemotherapy were firstly performed to screen out patients who were sensitive to chemotherapy. These patients were then infused with oxaliplatin via the superior rectal artery and oral capecitabine, combined with anti-PD1 antibody therapy for 2 cycles, and then underwent TME surgery. The primary endpoint of the study was the pCR rate.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed rectal adenocarcinoma
* Age ≥18 years old and ≤75 years old
* MRI stage T3-4aNany and TanyN1-2, but not T4b and no distant metastasis
* Life expectancy of 1 year The above
* Informed consent, no contraindications to chemotherapy exist
* The distance from the lower edge of the tumor to the anus is between 5cm to 12cm by MRI

Exclusion Criteria:

* Refused to participate in this study
* Multifocal colorectal cancer
* Past history of malignant tumors, except for basal cell carcinoma/papillary thyroid carcinoma/various types of carcinoma in situ
* Unable to receive chemotherapy , such as but not limited to bone marrow suppression, etc
* Major organ diseases (such as but not limited to COPD, coronary heart disease and renal insufficiency, etc.) acute attack and or severe acute infectious diseases (such as but not limited to hepatitis, pneumonia and myocarditis, etc.), ASA score> 3
* Mental disorder or illiteracy or language and communication barriers cannot understand the research plan
* There are contraindications to arterial puncture, such as but not limited to severe arteriosclerosis or even atresia, coagulation dysfunction, long-term use of anticoagulant drugs and cannot be stopped, etc
* Rectal tumor has obstruction or high risk of obstruction and or there is bleeding and/or perforation
* Peripheral sensory nerve disorder, unable to receive oxaliplatin chemotherapy
* Lateral pelvic lymph node metastasis (mainly supplied by internal iliac artery)
* Pregnancy or breastfeeding
* Unable to accept MRI examination
* Consecutive use of glucocorticoids for more than 3 days within 1 month before signing the consent form
* Tumor directly invades or adheres to adjacent organs、structures(T4b) or tumor invaded MRF（Mesoretal Fascia）
* Other scenarios deemed inappropriate by the investigators

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2024-04-25 (Estimated); Study Completion 2025-04-25 (Estimated)

PRIMARY OUTCOMES:
pCR rate | 1 day of postoperative pathological examination.
  the pathological complete remission rate of the rectal carcinoma

SECONDARY OUTCOMES:
DFS | From date of first chemotherapy until the date of first documented recurrence of tumor or date of death from any cause，whichever came first，assessed up to 36 months.
  3-year Disease-free survival
AE | From date of first chemotherapy until the date of patients were discharged from hospital after receiving TME operation, up to 20 weeks
  the rate of adverse event（AE）
Surgical Complication | within 30 days since operation
  the rate of surgical complication during or after operation
low anterior resection syndrome score | 3 months after operation; 6 months after operation;12 months after operation
  Low anterior resection syndrome (LARS) score of different time during treatment. The range (0-42) was divided into 0 to 20 (no LARS), 21 to 29 (minor LARS), and 30 to 42 (major LARS).
Concentration of FLT3LG | blood test of FLT3LG at baseline , pre-intervention of neoadjuvant chemotherapy, pre-intervention of artery infusion chemotherapy and pre-surgery.
  Fms Related Receptor Tyrosine Kinase 3 Ligand is a marker of immunogenic cell death
Concentration of cytokines | blood test of cytokines at baseline , pre-intervention of neoadjuvant chemotherapy, pre-intervention of artery infusion chemotherapy and pre-surgery.
  blood density measurement of immunoreaction associated cytokines
Concentration of DAMP | blood test of DAMP at baseline , pre-intervention of neoadjuvant chemotherapy, pre-intervention of artery infusion chemotherapy and pre-surgery.
  blood density measurement of damage-associated molecular pattern（DAMP）

CONTACTS AND LOCATIONS:
Overall Officials: Jun Li, MD, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No